CLINICAL TRIAL: NCT00558181
Title: Phase II Study of High-dose Methylprednisolone and Rituximab in Previously Treated Patients With High Risk Chronic B Lymphocytic Leukemia
Brief Title: High-dose Methylprednisolone and Rituximab in High Risk B-CLL
Acronym: LT-CLL-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Laimonas Griskevicius, Vilnius University Hospital Santariskiu Clinics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-CLL-001
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Chronic B-Lymphocytic Leukemia
Keywords: B CLL; Chronic B Lymphocytic Leukemia; Methylprednisolone; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — Rituximab; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab, Methylprednisolone (Experimental)
  Interventions: Drug: rituximab, methylprednisolone

INTERVENTIONS:
Drug: rituximab, methylprednisolone — Subjects will receive up-to 6 courses of IV infusion of Methylprednisolone and Rituximab every 21 day.

SUMMARY:
Studies have shown that both high-dose Methylprednisolone and Rituximab used as single agents are effective in relapsed and refractory B-CLL. Methylprednisolone acts independently of p53 apoptosis pathway. The combination of both drugs may improve response and outcome in previously treated high-risk B-CLL patients.

Study Objectives

Primary:

To determine the clinical benefit of high-dose Methylprednisolone and Rituximab in previously treated high-risk B-CLL patients in terms of clinical and flowcytometric response rate.

Secondary:

To determine progression free and overall survival. To characterize the safety profile of high-dose Methylprednisolone and Rituximab.

DETAILED DESCRIPTION:
Studies have shown that both high-dose Methylprednisolone and Rituximab used as single agents are effective in relapsed and refractory B-CLL. Methylprednisolone acts independently of p53 apoptosis pathway. The combination of both drugs may improve response and outcome in previously treated high-risk B-CLL patients.

Study Objectives

Primary:

To determine the clinical benefit of high-dose Methylprednisolone and Rituximab in previously treated high-risk B-CLL patients in terms of clinical and flowcytometric response rate.

Secondary:

To determine progression free and overall survival. To characterize the safety profile of high-dose Methylprednisolone and Rituximab.

Patient Population Patients with previously treated symptomatic high risk B-CLL 18 years of age and older.

Study Duration The study period for each subject is expected to be 21 months. Subjects will receive up-to 6 cycles of IV infusion of Methylprednisolone and Rituximab. Maximum duration of treatment is expected to be 9 months. All infusions of study treatment will be administered by medically qualified site staff in an inpatient or outpatient clinic under the supervision of an Investigator. Subjects will complete scheduled visits not later than Study Month 21, after which time they will enter into the long term follow up period. Subjects will be followed every 3 months for disease progression, initiation of subsequent leukemia treatment or survival, except in cases lost to follow up, or if a subject withdraws informed consent.

Study Design Phase II, multicenter, non-randomized, open label study.

Maximum Recruitment Period 2 years

Number of Planned Subjects Approximately 50 patients.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of CD20 positive chronic B lymphocytic leukemia (B-CLL) confirmed by biopsy or flow-cytometry.
2. Relapsed or progressive disease after at least 1 prior chemotherapy.
3. Stage Rai I-IV and progressive disease (according to NCI criteria). NCI progressive disease criteria16

Active B-CLL is defined by at least one of the following:

At least one of the disease related symptoms:

1. Constitutional symptoms:

   * Weight loss more 10 percent within the previous 6 months;
   * Fatigue (e. g. WHO performance status 2 or more);
   * Fever 38C or more 2 weeks or more without evidence of infection;
   * Night sweats without evidence of infection.
2. Evidence of progressive marrow failure as manifested by:

   * anemia (less 110 g/l) and / or
   * thrombocytopenia (less 100 x 109/l) within the previous 6 months and / or
   * neutropenia (less 1 x 109/l) within the previous 6 months.
3. Autoimmune hemolysis and / or thrombocytopenia poorly responsive to corticosteroid therapy.
4. Massive (i. e.6 cm or more bellow left costal margin) or progressive splenomegaly with progressive increase on 2 consecutive visits at least 2 weeks apart.
5. Massive lymphadenopathy or conglomerates (i.e., 10 cm or more in largest diameter) or progressive lymphadenopathy with increase on 2 consecutive visits at least 2 weeks apart.
6. Progressive lymphocytosis with an increase more 50 percent over a 2-month period or an anticipated doubling time of less than 6 months.

Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for protocol therapy

1. High-risk B-CLL biologically or clinically:

* Biologically high-risk B-CLL is defined by the presence of at least one of the following factors:
* 98 percent or more lgVH genes are homologous to the embryonic sequence and / or
* 17p del confirmed by FISH or
* 11q del confirmed by FISH or
* 12 trisomy.
* Clinically high-risk B-CLL is defined by the presence of at least one of the following factors:

  * Progressive or stable disease while on Fludarabine treatment.
  * Relapse after Fludarabine treatment within 12 months.
  * Older than 18 years.
  * Signed informed consent form.

Exclusion Criteria:

1. Intolerance to exogenous protein or known severe reaction to the administration of Rituximab.
2. Active infection.
3. Cancer radiotherapy, biological therapy or chemotherapy within 3 weeks prior to Study Day 1.
4. TBC or fungal infection within the past 6 months even if adequately controlled by treatment.
5. Severe organ deficiency preventing the participation in the study.
6. Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1.
7. Severe liver disease (total bilirubin or transaminases more 3 times ULN), except caused by the B-CLL.
8. Active peptic ulcer.
9. Inadequately controlled diabetes mellitus.
10. Suspected or confirmed B-CLL CNS disease.
11. Known to be HIV positive.
12. Difficult to control, uncooperative patients.
13. Allergic disorders in need of chronic glucocorticoid therapy.
14. Other oncological diseases requiring active treatment (except hormonal therapy).
15. Pregnancy and breastfeeding.
16. Patients of reproductive potential who are not using effective methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the ORR defined as the proportion of patients achieving CR, CR with MRD negativity (Complete Flow Cytometric Remission), nPR and PR. | End of treatment.

SECONDARY OUTCOMES:
PFS defined as time from the first day of treatment to the day the subject progresses or dies of any cause. OS defined as time from the first day of treatment to the day the subject dies of any cause. | End of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laimonas Griskevicius, PhD, MD, Principal Investigator — Vilnius University
Locations (2):
- Lithuania (2):
  - Klaipeda Seamen's Hospital, Klaipėda, Klaipėda County
  - Vilnius University Hospital Santariskiu Clinics, Vilnius, Vilnius County